CLINICAL TRIAL: NCT00216671
Title: Early Versus Late Initiation of Treatment With Risperdal Consta in Subjects With Schizophrenia After an Acute Episode
Brief Title: Long-acting Injectable Risperidone in Patients With Schizophrenia After an Acute Episode
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR002257
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2011-12-02 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; intramuscular injection; antipsychotic agents; long-acting risperidone
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 001 (Experimental): early initiation of treatment with Risperdal Consta 25 mg to 50 mg Risperdal Consta intrmuscular injection every 14 days starting at baseline. Treatment with oral antipsychotics or risperidone will continue 21 days after the first injection of Risperdal Consta. This treatment will then be tapered off within the next 7 days.
  Interventions: Drug: early initiation of treatment with Risperdal Consta
- 002 (Active Comparator): routine initiation of treatment with Risperdal Consta 25 mg to 50 mg Risperdal Consta intrmuscular injection every 14 days starting at week 12. Treatment with oral antipsychotics or risperidone will continue 21 days after the first injection of Risperdal Consta. This treatment will then be tapered off within the next 7 days.
  Interventions: Drug: routine initiation of treatment with Risperdal Consta

INTERVENTIONS:
Drug: early initiation of treatment with Risperdal Consta — 25 mg to 50 mg Risperdal Consta intrmuscular injection every 14 days starting at baseline. Treatment with oral antipsychotics or risperidone will continue 21 days after the first injection of Risperdal Consta. This treatment will then be tapered off within the next 7 days.
  Arms: 001
Drug: routine initiation of treatment with Risperdal Consta — 25 mg to 50 mg Risperdal Consta intrmuscular injection every 14 days starting at week 12. Treatment with oral antipsychotics or risperidone will continue 21 days after the first injection of Risperdal Consta. This treatment will then be tapered off within the next 7 days.
  Arms: 002

SUMMARY:
The primary objective of this randomized trial was to investigate whether early initiation of treatment with Risperdal Consta after an acute episode was not inferior to the routine approach (oral treatment for 12 weeks followed by treatment with Risperdal Consta). .

DETAILED DESCRIPTION:
Although many schizophrenia patients currently take oral antipsychotic medications, it is estimated that up to 75% of them have difficulty adhering to the daily oral regiment. Long-acting injectable formulations may eliminate the need for daily medication and enhance patient compliance with the treatment regimen. Traditionally, patients experiencing an episode of schizophrenia are first treated with oral medications until they are stabilized, and then injectable long-acting formulations are given. This is an open, multicenter, randomized Phase IV trial in patients after an acute episode of schizophrenia. Patients will be in the trial for 6 months. One treatment group will receive injections starting at baseline (early initiation); the other group will start with treatment as usual at baseline and begin injections at Week 12 (late initiation). Assessment of effectiveness include Positive And Negative Syndrome Scale (PANSS), in order to measure symptoms of schizophrenia; Clinical Global Impression - Severity (CGI-S), measuring overall severity of illness; Global Assessment of Functioning (GAF), assessesing overall psychological, social, and occupational functioning; and Quality of Life Questionnaire SF-12, measuring overall health status. Safety evaluations include the Extrapyramidal Symptoms Rating Scale (ESRS), incidence of adverse events throughout the study, and vital signs (pulse, blood pressure). The study hypothesis is that early initiation of long-acting risperidone injections is not inferior to late initiation as measured by changes in PANSS total score from baseline through endpoint (after 6 months). Risperidone, long-acting formulation for intramuscular injections (25 to 50 mg (maximum)), given every 14 days through 6 months, starting at baseline or Month 3. Treatment as usual for 3 months for late initiation group

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia by criteria of Diagnostic and Statistical Manual of Mental Diseases, Fourth Edition (DSM-IV)
* acute episode of schizophrenia within 2 weeks of study entry
* o subjects currently not treated or treated with oral antipsychotics or short-acting injectable antipsychotics (zuclopenthixol acutard is allowed) at doses not exceeding the registered dose
* Positive And Negative Syndrome Scale (PANSS) score >=80
* Clinical Global Impression - Severity (CGI-S) score >=5

Exclusion Criteria:

* DSM-IV axis I diagnosis other than schizophrenia
* known hypersensitivity or lack of response to risperidone
* pregnant or nursing females, or those without adequate contraception
* alcohol or drug abuse or dependence diagnosed in the last month prior to entry,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2005-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.
Locations (31):
- Denmark (4):
  - Copenhagen
  - Glostrup Municipality
  - Hjørring
  - Kolding
- Finland (2):
  - Helsinki
  - Vantaa
- France (6):
  - Bar-le-Duc
  - Beaupuy
  - Clermont-Ferrand
  - Colmar
  - La Seyne-sur-Mer
  - Mont-Saint-Martin
- Greece (4):
  - Athens
  - Chania
  - Thessalonikis
  - Tripoli
- Israel (3):
  - Bat Yam
  - Pardesiyya
  - Petah Tikva
- Levanger, Norway
- Ljubljana, Slovenia
- Sweden (5):
  - Danderyd
  - Gothenburg
  - Huddinge
  - Stockholm
  - Trollhättan
- Switzerland (3):
  - Oetwil
  - Sankt Urban
  - Zurich
- United Kingdom (2):
  - London
  - Norfolk

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Initiation of Treatment: 25 mg to 50 mg Risperdal Consta intramuscular (i.m.) injection every 14 days starting at baseline. Treatment with oral antipsychotics (APs) or risperidone will continue 21 days after the first injection of Risperdal Consta. This treatment will then be tapered off within the next 7 days.
- Late Initiation of Treatment: routine practice: The oral AP treatment started during the acute episode will be maintained until week 12. Starting at week 12, 25 mg to 50 mg Risperdal Consta i.m. injection every 14 days. Treatment with previous oral APs will continue 21 days after the first injection and then be tapered off within the next 7 days.
Period: Overall Study
Arm/Group | Early Initiation of Treatment | Late Initiation of Treatment
Started | 110 | 110
Completed | 75 | 60
Not Completed | 35 | 50
Not completed — Adverse Event | 4 | 9
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Refused Injections | 3 | 13
Not completed — No Need to Continue Medication | 1 | 1
Not completed — Insufficient Response | 9 | 4
Not completed — Lost to Follow-up | 3 | 5
Not completed — Non compliant | 2 | 2
Not completed — Ineligible | 0 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Protocol Violation | 3 | 5
Not completed — Relapse | 1 | 0
Not completed — Investigator Illness | 0 | 1
Not completed — Patient Moved | 0 | 1
Not completed — Ineligible, no efficacy data | 2 | 2
Not completed — Insufficient Response Adverse Event | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Early Initiation of Treatment: 25 mg to 50 mg Risperdal Consta intramuscular (i.m.) injection every 14 days starting at baseline. Treatment with oral antipsychotics (APs) or risperidone will continue 21 days after the first injection of Risperdal Consta. This treatment will then be tapered off within the next 7 days. Two enrolled patients were excluded from the baseline analysis as these patients dropped out early and no safety or efficacy data were present.
- Late Initiation of Treatment: routine practice: The oral AP treatment started during the acute episode will be maintained until week 12. Starting at week 12, 25 mg to 50 mg Risperdal Consta i.m. injection every 14 days. Treatment with previous oral APs will continue 21 days after the first injection and then be tapered off within the next 7 days. Two enrolled patients were excluded from the baseline analysis as these patients dropped out early and no efficacy data were present.
- Total: Total of all reporting groups
Arm/Group | Early Initiation of Treatment | Late Initiation of Treatment | Total
Number analyzed (Participants) | 108 | 108 | 216
Age Continuous [Mean (Standard Deviation); unit: years] — Two enrolled patients from each group were excluded from the baseline analysis as these patients dropped out early and no safety or efficacy data were present.
  years | 38 (11) | 38 (11) | 38 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 43 | 84
  Male | 67 | 65 | 132

OUTCOME MEASURES:

1. Primary Outcome: Change in Positive And Negative Syndrome Scale (PANSS) Total Score From Baseline to Endpoint
Description: The PANSS is a specific scale for the measurement of the symptoms of schizophrenia. Symptoms of schizophrenia will be assessed using the 30-item PANSS scale. Each item of the scale is to be scored on a scale of 1 (absent) to 7 (extreme).The total score can range from 30 to 210.
Time Frame: at baseline and Week 26 or at premature discontinuation
Population: Per Protocol analysis: all randomized patients who had no violation on eligibility criteria or no major protocol violation. This excluded 42 patients in the early and 34 in the late initiation group. 1 patient in the early initiation group had no PANSS at endpoint. The endpoint is the last post-baseline value of the patient.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Early Initiation of Treatment | Late Initiation of Treatment
Number analyzed (Participants) | 65 | 74
scores on a scale | -38.37 (23.1) | -37.24 (25.02)
Statistical Analysis 1: Comparison: Early Initiation of Treatment vs Late Initiation of Treatment; Assuming a difference of 3 points in favor of early initiation of treatment with Risperdal Consta, a sample size of 87 subjects per treatment arm has a power of 80% to demonstrate non-inferiority at the 0.025-level (1-sided). It was expected that about 20% of randomized subjects had to be excluded from the per-protocol (PP) analysis. Therefore, 220 subjects were to be included; Test type: Non-Inferiority or Equivalence — Non-inferiority of early initiation was inferred if the upper 95% confidence boundary for the difference of change in PANSS total score from baseline in favor of the routine approach is less than 6; p = 0.784, ANCOVA — An ANCOVA model with treatment as factor was used. The comparison between the 2 treatment groups was performed based on the least-squares means obtained from the ANCOVA model; Mean Difference (Net) = -1.13, 95% CI 2-sided [-9.24 to 6.99], Standard Error of Mean 4.10

2. Secondary Outcome: Change From Baseline in PANSS Total Score at Week 6
Description: The PANSS is a specific scale for the measurement of the symptoms of schizophrenia. Symptoms of schizophrenia will be assessed using the 30-item PANSS scale. Each item of the scale is to be scored on a scale of 1 (absent) to 7 (extreme). The total score can range from 30 to 210.
Time Frame: at baseline and Week 6.
Population: Per protocol population. This excluded 42 patients in the early start group and 34 patients in the late start group. An additional 3 and 5 patients in the respective groups had missing PANSS data at week 6.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Early Initiation of Treatment | Late Initiation of Treatment
Number analyzed (Participants) | 63 | 69
scores on a scale | -27.48 (17.97) | -27.96 (20.10)

3. Secondary Outcome: Change From Baseline in PANSS Total Score at Week 12
Description: as for outcome 2
Time Frame: at baseline and Week 12.
Population: Per protocol population. This excluded 42 patients in the early start group and 34 patients in the late start group. An additional 9 and 23 patients in the respective groups had missing PANSS data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Early Initiation of Treatment | Late Initiation of Treatment
Number analyzed (Participants) | 57 | 51
scores on a scale | -35.84 (22.83) | -34.49 (19.12)

4. Secondary Outcome: Change From Baseline to Endpoint in Clinical Global Impression - Severity (CGI-S)
Description: The CGI-S rating scale is used to rate the severity of a subject's psychotic condition on a 7-point scale ranging from 1 (not ill) to 7 (extremely severe). This scale permits a global evaluation of the subject's condition at a given time.
Time Frame: at baseline and endpoint (week 26 or at premature discontinuation).
Population: Per protocol population. This excluded 42 patients in the early start group and 34 patients in the late start group.One additional patient in the Early Initiation group has missing CGI-S data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Early Initiation of Treatment | Late Initiation of Treatment
Number analyzed (Participants) | 65 | 74
scores on a scale | -1.91 (1.35) | -2.03 (1.27)
Statistical Analysis 1: Comparison: Early Initiation of Treatment vs Late Initiation of Treatment; Between-group comparison of the change in CGI-S from baseline to endpoint was analyzed as is with no derived calculations. CGI-S scores were coded as follows: 0=normal, not at all ill, 1=borderline, etc. and 6=among the most extremely ill patients.The endpoint of the study was based on the Last Observation Carried Forward (LOCF) principle, i.e., it was defined as the last available visit during the study with non-missing data for a parameter (excluding the baseline value); Test type: Superiority or Other; p = 0.800, Wilcoxon two sample test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 2: Comparison: Early Initiation of Treatment; Within-group comparison of the change in CGI-S from baseline to endpoint was analyzed as is with no derived calculations. CGI-S scores were coded as follows: 0=normal, not at all ill, 1=borderline, etc. and 6=among the most extremely ill patients; Test type: Superiority or Other; p < 0.001, Wilcoxon-signed-rank test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 3: Comparison: Late Initiation of Treatment; [analysis description as in outcome 4, analysis 2]; Test type: Superiority or Other; p < 0.001, Wilcoxon-signed-rank test — The statistical test was interpreted at the 5% significance level

5. Secondary Outcome: Change From Baseline to Endpoint in Global Assessment of Functioning (GAF)
Description: Overall psychological, social, and occupational functioning is rated on a scale of mental health-illness from 1 being the worst functioning to 100 being the best. Impairment in functioning due to physical (or environmental) limitations must not be included in the rating.
Time Frame: at baseline and endpoint (week 26 or at premature discontinuation).
Population: Per protocol population. This excluded 42 patients in the early start group and 34 patients in the late start group.One additional patient in the Early Initation group has missing GAF data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Early Initiation of Treatment | Late Initiation of Treatment
Number analyzed (Participants) | 65 | 74
scores on a scale | 19.65 (14.20) | 18.72 (16.76)
Statistical Analysis 1: Comparison: Early Initiation of Treatment vs Late Initiation of Treatment; Between-group comparison of the change in GAF from baseline to endpoint. The endpoint of the study was based on the Last Observation Carried Forward (LOCF) principle, i.e., it was defined as the last available visit during the study with non-missing data for a parameter (excluding the baseline value); Test type: Superiority or Other; p = 0.798, Wilcoxon two sample test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 2: Comparison: Early Initiation of Treatment; Within-group comparison of the change in GAF from baseline to endpoint. The endpoint of the study was based on the Last Observation Carried Forward (LOCF) principle, i.e., it was defined as the last available visit during the study with non-missing data for a parameter (excluding the baseline value); Test type: Superiority or Other; p < 0.001, Wilcoxon-signed-rank test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 3: Comparison: Late Initiation of Treatment; [analysis description as in outcome 5, analysis 2]; Test type: Superiority or Other; p < 0.001, Wilcoxon-signed-rank test — The statistical test was interpreted at the 5% significance level

6. Secondary Outcome: Change From Baseline to Endpoint in Quality of Life Questionnaire SF-12
Description: Short Form Health Survey: A generic dual-ie, mental and physical health-scale measure of quality of life. This is a 12-item subset of the SF-36 survey that measures the same 8 domains of health. As a brief, reliable measure of overall health status, the SF-12 is the instrument of choice in large population health surveys and has been used extensively as a screening tool. SF-12 will be filled in by the patient. The scores range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Time Frame: at baseline, Weeks 6, 12, and endpoint (week 26 or at premature discontinuation).
Population: Per protocol population. This excluded 42 patients in the early start group and 34 patients in the late start group.An additional 9 and 11 patients in the respective groups had missing SF-12 data.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Early Initiation of Treatment | Late Initiation of Treatment
Number analyzed (Participants) | 57 | 63
scores on a scale
  Physical Component Summary (PCS) | 2.76 (10.73) | 1.75 (7.93)
  Mental Component Summary (MCS) | 3.25 (9.19) | 2.96 (10.76)
Statistical Analysis 1: Comparison: Early Initiation of Treatment vs Late Initiation of Treatment; Between-group comparison of the change in SF-12 PCS score from baseline to endpoint. The endpoint of the study was based on the Last Observation Carried Forward (LOCF) principle, i.e., it was defined as the last available visit during the study with non-missing data for a parameter (excluding the baseline value); Test type: Superiority or Other; p = 0.519, Wilcoxon two sample test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 2: Comparison: Early Initiation of Treatment; Within-group comparison of the change in SF-12 PCS score from baseline to endpoint. The endpoint of the study was based on the Last Observation Carried Forward (LOCF) principle, i.e., it was defined as the last available visit during the study with non-missing data for a parameter (excluding the baseline value); Test type: Superiority or Other; p < 0.001, Wilcoxon-signed-rank test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 3: Comparison: Late Initiation of Treatment; [analysis description as in outcome 6, analysis 2]; Test type: Superiority or Other; p < 0.001, Wilcoxon-signed-rank test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 4: Comparison: Early Initiation of Treatment vs Late Initiation of Treatment; Between-group comparison of the change in SF-12 MCS score from baseline to endpoint. The endpoint of the study was based on the Last Observation Carried Forward (LOCF) principle, i.e., it was defined as the last available visit during the study with non-missing data for a parameter (excluding the baseline value); Test type: Superiority or Other; p = 0.721, Wilcoxon two sample test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 5: Comparison: Early Initiation of Treatment; Within-group comparison of the change in SF-12 MCS score from baseline to endpoint. The endpoint of the study was based on the Last Observation Carried Forward (LOCF) principle, i.e., it was defined as the last available visit during the study with non-missing data for a parameter (excluding the baseline value); Test type: Superiority or Other; p < 0.001, Wilcoxon-signed-rank test — The statistical test was interpreted at the 5% significance level
Statistical Analysis 6: Comparison: Late Initiation of Treatment; [analysis description as in outcome 6, analysis 5]; Test type: Superiority or Other; p < 0.001, Wilcoxon-signed-rank test — The statistical test was interpreted at the 5% significance level

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring between the first study-related procedure, i.e. screening visit, and week 26 or early termination were reported.
Description: AEs described hereafter are treatment-emergent AEs, defined as AEs that were new in onset or aggravated in severity following treatment start.
Arm/Group | Early Initiation of Treatment | Late Initiation of Treatment
Serious Adverse Events (participants affected / at risk) | 18/110 | 22/110
Other Adverse Events (participants affected / at risk) | 58/110 | 66/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Initiation of Treatment (N=110) | Late Initiation of Treatment (N=110)
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Drug Toxicity (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 2 | 2
Dizziness (Nervous system disorders) | 0 | 1
Extrapyramidal Disorder (Nervous system disorders) | 3 | 0
Mental Impairment (Nervous system disorders) | 0 | 1
Neuroleptic Malignant Syndrome (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Acute Psychosis (Psychiatric disorders) | 1 | 0
Aggression (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 4 | 4
Delusion (Psychiatric disorders) | 1 | 1
Depressed Mood (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 0 | 1
Hallucination (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 2
Psychiatric Symptom (Psychiatric disorders) | 0 | 1
Psychotic Disorder (Psychiatric disorders) | 2 | 1
Schizophrenia (Psychiatric disorders) | 3 | 5
Schizophrenia, Paranoid Type (Psychiatric disorders) | 1 | 3
Suicidal Ideation (Psychiatric disorders) | 0 | 3
Urinary Incontinence (Renal and urinary disorders) | 0 | 1
Epididymitis (Reproductive system and breast disorders) | 1 | 0
Erysipelas (Skin and subcutaneous tissue disorders) | 1 | 0
Self-medication (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Early Initiation of Treatment (N=110) | Late Initiation of Treatment (N=110)
Asthenia (General disorders) | 1 | 4
Weight Increased (Investigations) | 8 | 8
Akathisia (Nervous system disorders) | 8 | 7
Dystonia (Nervous system disorders) | 4 | 0
Extrapyramidal Disorder (Nervous system disorders) | 3 | 9
Headache (Nervous system disorders) | 3 | 5
Sedation (Nervous system disorders) | 2 | 7
Somnolence (Nervous system disorders) | 1 | 5
Tremor (Nervous system disorders) | 6 | 3
Anxiety (Psychiatric disorders) | 5 | 6
Depression (Psychiatric disorders) | 5 | 5
Insomnia (Psychiatric disorders) | 9 | 10
Erectile Dysfunction (Reproductive system and breast disorders) | 2 | 5
Hypertension (Vascular disorders) | 3 | 1
Tension (Psychiatric disorders) | 3 | 2
Aggression (Psychiatric disorders) | 3 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Tootache (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
Due to the substantial number of protocol deviations (mainly due to prohibited medication), the study did not have the required power to demonstrate non-inferiority in the per protocol population

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days